CLINICAL TRIAL: NCT07203339
Title: Home-based Transcranial Direct Current Stimulation (tDCS) Compared to Duloxetine in the Treatment of Fibromyalgia: a Randomized Non-inferiority Clinical Trial (FIBROSTIM)
Brief Title: Home-based Transcranial Direct Current Stimulation (tDCS) Compared to Duloxetine: Non-inferiority Clinical Trial (FIBROSTIM)
Acronym: FIBROSTIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 85778525.8.0000.5327
Record Dates: First submitted 2025-06-04; First posted 2025-10-02 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Fibromyalgia (FM); tDCS; Duloxetine; BDNF; EEG
Keywords: Fibromyalgia; Transcranial Direct Current Stimulation; Duloxetine; Biomarkers; Precision Medicine
MeSH Terms: conditions — Fibromyalgia | interventions — Transcranial Direct Current Stimulation; Duloxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Arm 1: Duloxetine + Sham tDCS (n = 244) Duloxetine 60 mg/day plus 28 sessions of sham tDCS (30s stimulation at start, 10 min, and end), with electrodes placed over left M1 (anode) and right supraorbital area (cathode), using 35 cm² electrodes. Sessions are home-based, 20 minutes/day for 4 weeks.
  Arm 2: Active tDCS + Placebo (n = 244) Active tDCS (2 mA, 20 minutes/day for 4 weeks) using the same montage, plus oral placebo. Sessions are home-based following in-person training. The device monitors contact impedance and logs session data.
  Arm 3: Sham tDCS + Placebo (n = 122) Sham tDCS and oral placebo, using the same procedures as above.
  Common to all arms:
  All participants receive home-based physical exercise guidance and pain neuroscience education. Duloxetine and matching placebo (30 mg and 60 mg) are prepared and labeled by a compounding pharmacy using a double-dummy design. Medication kits follow a titration and tapering schedule and are dispensed at study visits.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Researchers will receive a tDCS device pre-programmed by biomedical engineering, without prior knowledge of whether the condition is active or sham.
  The compounding pharmacy contracted for the study will prepare the placebo and fractionate the Duloxetine Hydrochloride. Researchers will receive a kit containing four labeled containers:
  Containers 1 and 4 (white lid): 7 capsules of either placebo or Duloxetine 30 mg
  Container 2 (green lid): 16 capsules of either placebo or Duloxetine 60 mg
  Container 3 (green lid): 42 capsules of either placebo or Duloxetine 60 mg
  Each container will display the randomization ID and will be properly labeled. Allocation information will be accessible only to the responsible pharmacist (who is not involved in data collection) and the researcher who performed the randomization (with no contact with participants). Labels will include the project number (CAAE), participant ID (RedCap), and pharmacist's name.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- (s-tDCS over M1+placebo medication) - Home-Based Transcranial Direct Current Stimulation (tDCS) (Sham Comparator): The sham tDCS protocol will use the same electrode montage as the active tDCS, with active current delivered for 30 seconds at the beginning, after 10 minutes, and at the end of the session. The current will be applied using 35 cm² electrodes.
  Interventions: Device: Transcranial direct current stimulation (tDCS) plus placebo.; Device: Home-based transcranial direct current stimulation
- The study includes 28 sessions of home-based anodal transcranial direct current stimulation (tDCS) (Experimental): Active anodal tDCS (2 mA) or sham tDCS will be applied over the left M1 (anode) and the right supraorbital area (cathode) for 20 minutes, combined with physical exercises and educational guidance on pain neuroscience for fibromyalgia. After in-person training, participants will receive instructions for home use.
  Interventions: Device: Transcranial direct current stimulation (tDCS) plus placebo.; Device: Home-based transcranial direct current stimulation
- Duloxetine 60 mg (Active Comparator): The pharmacological intervention will use duloxetine (30 mg and 60 mg), commercially acquired. The medication and placebo will be sourced via contracts with a compounding pharmacy and a retail drugstore. Generic Duloxetine Hydrochloride (Germed) will be purchased and sent for fractioning and placebo preparation.
  Each participant will receive a kit with four jars (duloxetine or placebo):
  Jar 01 (white lid): 7 × 30 mg - Week 1 (run-in); Jar 02 (green lid): 16 × 60 mg - Weeks 2-3 (run-in); Jar 03 (green lid): 42 × 60 mg - During tDCS; Jar 04 (white lid): 7 × 30 mg - Post-treatment taper.
  Interventions: Drug: Duloxetine (60 mg) once daily; Drug: Duloxetine 60 mg

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) plus placebo. — Participants will be randomized to receive 28 sessions of active anodal tDCS (2 mA) or sham, with the anode over the left M1 and the cathode over the right supraorbital area, for 20 minutes, combined with pain neuroscience education and physical exercises. Sessions will be self-administered at home, daily for 4 weeks. Electrodes (35 cm²) will be placed using neoprene caps (sizes S to XL), adjusted according to head circumference. Monitoring: the device records session time, duration, and adherence, interrupting the session if impedance exceeds 1 mA (5-second interval) or if current varies >10%. Developed in partnership with HCPA's Biomedical Engineering, the device is licensed by UFRGS/HCPA and registered with ANVISA (No. 80079190028).
  Arms: (s-tDCS over M1+placebo medication) - Home-Based Transcranial Direct Current Stimulation (tDCS); The study includes 28 sessions of home-based anodal transcranial direct current stimulation (tDCS)
Drug: Duloxetine (60 mg) once daily — Duloxetine (30 mg and 60 mg) will be purchased from a commercial pharmacy and fractionated by a compounding pharmacy, which will also prepare the placebo. Capsules will be transferred into standardized jars based on dosing schedule:
  * Jar 01 (white cap): 7 capsules of 30 mg
  * Jar 02 (green cap): 16 capsules of 60 mg
  * Jar 03 (green cap): 42 capsules of 60 mg
  * Jar 04 (white cap): 7 capsules of 30 mg Placebo and duloxetine capsules will be identical in appearance. Kits will be labeled with CAEE number, participant ID (RedCap), pharmacist and PI names, and storage/use instructions. Kits will be stored at the HCPA Pharmacy Service under controlled conditions and dispensed during visits AV1 (Jars 1 and 2), AV2 (Jar 3), and AV3 (Jar 4).
  Arms: Duloxetine 60 mg
Device: Home-based transcranial direct current stimulation — Participants will be randomized to receive 28 sessions of active anodal tDCS (2 mA) anode over the left M1 and the cathode over the right supraorbital area, for 20 minutes
  Arms: (s-tDCS over M1+placebo medication) - Home-Based Transcranial Direct Current Stimulation (tDCS); The study includes 28 sessions of home-based anodal transcranial direct current stimulation (tDCS)
Drug: Duloxetine 60 mg — Duloxetine (30 mg and 60 mg) will be purchased from a commercial pharmacy and fractionated by a compounding pharmacy, which will also prepare the placebo. Capsules will be transferred into standardized jars based on dosing schedule:
  * Jar 01 (white cap): 7 capsules of 30 mg
  * Jar 02 (green cap): 16 capsules of 60 mg
  * Jar 03 (green cap): 42 capsules of 60 mg
  * Jar 04 (white cap): 7 capsules of 30 mg Placebo and duloxetine capsules will be identical in appearance. Kits will be labeled with CAEE number, participant ID (RedCap), pharmacist and PI names, and storage/use instructions. Kits will be stored at the HCPA Pharmacy Service under controlled conditions and dispensed during visits AV1 (Jars 1 and 2), AV2 (Jar 3), and AV3 (Jar 4).
  Arms: Duloxetine 60 mg

SUMMARY:
Fibromyalgia is characterized by widespread pain, fatigue, non-restorative sleep, and psychocognitive alterations, compromising quality of life and leading to absenteeism and early retirement. Up to 70% of patients discontinue treatment with antidepressants and anticonvulsants due to adverse effects or low efficacy, and more than 30% resort to opioid use. Given the treatment challenges and the scarcity of safe alternatives, there is growing interest in interventions such as transcranial direct current stimulation (tDCS), which has shown efficacy in improving symptoms and functionality, with low cost and few side effects. In this context, we designed a randomized, double-blind, double-dummy clinical trial to compare the non-inferiority of 28 home-based anodal tDCS (2 mA) applied over the primary motor cortex (M1) versus duloxetine 60 mg. Both treatments will be combined with physical exercise and pain education. Outcomes will be assessed through multidimensional measures of pain, functionality, global impression of improvement, and the function of the descending pain inhibitory system. Secondary outcomes include quality of life, depressive symptoms, psychophysical pain measures, and treatment adherence. An additional analysis will compare the results of sham tDCS and duloxetine placebo within the non-inferiority model. Predictors of treatment response will also be explored, including symptom severity and oscillatory patterns of cortical electrical activity, rest-activity rhythm, and autonomic function assessed by R-R interval. Furthermore, serum levels of S100-B protein, brain-derived neurotrophic factor (BDNF), and genetic variants related to neuroplasticity in the BDNF Val66Met, Catechol-O-Methyltransferase (COMT) (rs4680) (G>A), OPRM1, and PER2 genes will be analyzed. Inflammatory markers (TNF-α, IL-1, IL-2, IL-6, IL-10, C-reactive protein) and serum endorphins will also be assessed. A total of 610 women with fibromyalgia (aged 18 to 75 years) will be randomized into three groups (2:2:1): duloxetine + sham tDCS (n=244); active tDCS + placebo (n=244); and sham tDCS + placebo (n=122). Participants will be assessed during treatment and at 3, 6, and 12 months after completing the intervention protocol. An interim analysis will be conducted when ~50% of participants (n ≈ 305) complete the 3-month follow-up by an independent, blinded Data Monitoring Committee (DMC). (i) The trial may be stopped if the conditional probability of demonstrating non-inferiority is <10%, based on frequentist or Bayesian methods. (i) The trial will be stopped if serious adverse events (SAEs) in the active tDCS group increase by ≥30% compared to duloxetine (p < 0.01, adjusted). (ii) Early stopping for efficacy will be considered if active tDCS demonstrates clear non-inferiority or superiority over duloxetine on the primary outcome. Superiority requires: (iii) a clinically relevant difference exceeding the non-inferiority margin (≥10% pain reduction); (ii) statistical significance (p < 0.005, O'Brien-Fleming adjusted); and (iii) a ≥2-point (20%) improvement on the BPI, confirmed in the ITT analysis. This study aims to generate evidence to support the decision-making process of the National Committee for Health Technology Incorporation (CONITEC) regarding the availability of tDCS in the Brazilian Unified Health System (SUS). In addition, identifying predictors of response to tDCS and duloxetine, through the integration of genetic, neurophysiological, inflammatory, and psychosocial markers using machine learning algorithms, will allow for identifying factors that can personalize fibromyalgia treatment. This approach enhances clinical efficacy, reduces costs associated with ineffective interventions, and supports more accurate therapeutic decisions, expanding access to safe, effective, and sustainable care within the public healthcare system

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria:

* Woman aged between 18 and 75 years
* Right-handed
* Literate in reading and writing
* Clinical diagnosis of fibromyalgia based on the American College of Rheumatology (ACR) 2010-2016 criteria
* Numeric Pain Scale (NPS) score ≥ 4 on most days in the past 30 days
* Agree no changes in medication dosage during the treatment period (except for analgesics)
* Able to swallow tablets
* Able to understand instructions for using tDCS at home

Exclusion Criteria:

* Living more than 250 km from Porto Alegre
* Pregnancy
* Decompensated systemic diseases
* Chronic inflammatory rheumatologic diseases
* Untreated hypothyroidism
* Active cancer under treatment
* Alcohol or drug abuse in the past 6 months
* Decompensated psychiatric disorders with suicide risk and a defined plan
* Use of duloxetine at a dose > 60 mg/day
* Metal implants in the brain
* Implanted brain medical devices
* Cardiac pacemaker
* Cochlear implant
* Neurological disorders
* History of traumatic brain injury or neurosurgery

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Pain Interference | Participants will undergo weekly home-based assessments during both the run-in period (Weeks 1 to 3) and the treatment phase (Weeks 4 to 7), as well as at 3, 6, and 12 months after the end of the intervention
  The Brief Pain Inventory (BPI) assesses pain intensity and interference across seven domains, generating a global interference index using 0-10 scales.
Patient Global Impression of Improvement | To be assessed at Visit 4, after completing the four-week treatment with either active (a-tDCS), s-tDCS), or duloxetine
  Patient Global Impression of Improvement (PGI-I): A 7-point scale that assesses the patient's overall perception of change in their condition, ranging from 'very much worse' (1) to 'very much improved' (7). Higher scores indicate greater perceived improvement (e.g., reduced symptoms or better functioning), while lower scores reflect worsening of symptoms or condition.
Impact of fibromyalgia symptoms on quality of life | Participants will be assessed at Visit 1 (prior to the run-in period), at Visit 4 (after completing the four-week treatment with active [a-tDCS], sham [s-tDCS], or duloxetine), and again at 3, 6, and 12 months following the end of the treatment.
  Fibromyalgia Impact Questionnaire (FIQ): Brazilian version assessing quality of life across function, overall impact, and symptoms. Scores range from 0 to 100, with higher scores indicating greater impact of fibromyalgia on the individual's daily life and functioning.
Cognitive symptoms | Participants will be assessed at Visit 1 (before the run-in period), at Visit 4 (after completing the four-week treatment with active [a-tDCS], sham [s-tDCS], or duloxetine), and again at 3, 6, and 12 months after the end of the treatment.
  Barkley Deficits in Executive Functioning Scale (Short Form).Each item is rated on a Likert scale from 1 (never or rarely) to 4 (very often), resulting in a total score range of 20 to 80, with higher scores indicating greater executive functioning impairment
Function of the descending pain inhibitory system | Participants will be assessed at Visit 1 (before the run-in period) and at Visit 4 (after completing the four-week treatment with active [a-tDCS], sham [s-tDCS], or duloxetine).
  Conditioned Pain Modulation (CPM) test: This test assesses descending pain inhibition.
  This test assesses the efficiency of descending pain inhibitory pathways. Pain intensity is rated using a verbal numerical rating scale (0 = no pain to 10 = worst possible pain) before (T0) and during (T1) cold-water immersion. The CPM effect is calculated as the difference between pain ratings at T0 and T1, with greater reductions indicating more effective pain inhibition.
Cortical Electrical Activity | Participants will be assessed at Visit 1 (before the run-in period) and at Visit 4 (after completing the four-week treatment with active [a-tDCS], sham [s-tDCS], or duloxetine).
  Cortical electrical activity will be assessed using resting-state electroencephalography (EEG). Recordings will be performed in a quiet room, with participants seated comfortably and instructed to remain relaxed and still. EEG data will be collected during eyes-closed and eyes-open conditions using a 64-channel EEG system. Signals will be recorded with a band-pass filter of 0.3-200 Hz and a sampling rate of 250 Hz. Spectral power measures will be analyzed to characterize cortical oscillatory activity associated with pain processing and central sensitization in fibromyalgia.

SECONDARY OUTCOMES:
Depressive Symptoms | Assessment timepoints: Baseline; Week 8 (Visit 4/after completing the four-week treatment with active [a-tDCS], sham [s-tDCS], or duloxetine); 3 months post-treatment; 6 months post-treatment; 12 months post-treatment.
  Assessed using the Beck Depression Inventory-II (BDI-II), a 21-item self-report questionnaire with total scores ranging from 0 to 63. Higher scores indicate greater severity of depressive symptoms
Subjective Sleep Quality | Assessment timepoints: Baseline; Week 8 (Visit 4/after completing the four-week treatment with active [a-tDCS], sham [s-tDCS], or duloxetine); 3 months post-treatment; 6 months post-treatment; 12 months post-treatment.
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), a self-questionnaire that evaluates sleep quality over the past month. It generates a global score ranging from 0 to 21, with higher scores indicating poorer sleep quality.
Circadian Profile (Chronotype) | Assessment timepoints: Baseline; Week 8 (Visit 4/after completing the four-week treatment with active [a-tDCS], sham [s-tDCS], or duloxetine); 3 months post-treatment; 6 months post-treatment; 12 months post-treatment.
  Chronotype will be measured using the Munich ChronoType Questionnaire (MCTQ) which evaluates individual sleep-wake patterns and chronotype based on the timing of sleep on workdays and free days. The key metric is the mid-sleep point on free days (MSF), which is based on sleep onset and wake-up times. The corrected version (MSFsc) accounts for workweek sleep debt and better reflects chronotype: lower values indicate morning types; higher values, evening types.
Objective Sleep and Activity (Actigraphy) | Actigraph use during the run-in period (Weeks 1 to 3) and throughout the treatment phase (weeks 4 to 7)
  Actigraphy (accelerometer) assesses sleep quality and physical mobility. Mean values are calculated across days for parameters such as total sleep time, sleep efficiency, and activity levels. Higher sleep efficiency and activity indicate better sleep quality and physical functioning; lower values suggest disturbances or impairment.
Analgesic Use | Analgesic use during the run-in period (Weeks 1 to 3) and throughout the treatment phase (Weeks 4 to 7).
  The use of analgesics will be assessed by recording the number of tablets of each analgesic taken per week during the run-in period (Weeks 1 to 3) and throughout the treatment phase (Weeks 4 to 7)
Functional Capacity | Assessment timepoints: Baseline; Week 8 (Visit 4/after completing the four-week treatment with active [a-tDCS], sham [s-tDCS], or duloxetine); 3 months post-treatment; 6 months post-treatment; 12 months post-treatment.
  Functional interference of pain is assessed using the Brazilian Profile of Chronic Pain: Screen (B-PCP: S), which captures pain intensity, interference in daily life, and emotional impact. Scores range from 0 to 100, with higher scores indicating greater pain-related interference and effects.
Heat Pain Threshold | Assessment timepoints: Baseline; Week 8 (Visit 4/after completing the four-week treatment with active [a-tDCS], sham [s-tDCS], or duloxetine)
  Heat pain threshold will be assessed via quantitative sensory testing (QST) on the left forearm using a thermode that increases temperature from 30°C to 52°C at a rate of 1°C per second. The pain threshold is calculated as the average temperature at which pain is first reported across three trials. Higher values indicate greater pain threshold.
Pressure Pain Threshold | Assessment timepoints: Baseline; Week 8 (Visit 4/after completing the four-week treatment with active [a-tDCS], sham [s-tDCS], or duloxetine)
  Pressure pain threshold will be measured using a pressure algometer applied to the left forearm. The threshold is defined as the point at which pressure sensation becomes painful, averaged across three trials. Higher values indicate lower pain sensitivity.
Cold Pressor Test Pain Intensity | Assessment timepoints: Baseline; Week 8 (Visit 4/after completing the four-week treatment with active [a-tDCS], sham [s-tDCS], or duloxetine)
  Cold Pressor Test: Non-dominant hand immersed in ice water (~1°C) for up to 2 minutes with continuous movement. Pain intensity is continuously rated via electronic visual analog scale (0-100%), enabling calculation of peak pain, mean pain, and area under the curve (AUC).allowing calculation of peak pain, mean pain, and area under the curve (AUC). Higher scores reflect greater pain intensity.
Patient-Defined Goals | Assessment timepoints: Baseline; Week 8 (Visit 4/after completing the four-week treatment with active [a-tDCS], sham [s-tDCS], or duloxetine)
  Patients will select three priority areas-physical, psychological, functional, or social-and define personalized, measurable goals at Visit 1 (V1) and evaluate them at the end of the treatment period (Visit 4).
Treatment Adherence | Assessment timepoints: Week 8 (Visit 4/after completing the four-week treatment with active [a-tDCS], sham [s-tDCS], or duloxetine)
  tDCS adherence: Assessed by the number and duration of valid sessions recorded by the device software, based on impedance and resistance parameters.
  Pharmacological treatment adherence:
  Assessed by pill count at Visit 3 and Visit 4, based on the number of capsules consumed
Side Effects | Assessment timepoints: During the run-in period (Weeks 1 to 3) and throughout the treatment phase (Weeks 4 to 7).
  The adverse effects of duloxetine will be assessed weekly throughout the run-in period (Weeks 1 to 3) and during the treatment phase (Weeks 4 to 7) using structured questionnaires that include common side effects such as nausea, dry mouth, dizziness, and somnolence, which will be recorded as 'yes' or 'no'. Adverse effects related to tDCS-such as tingling, itching, burning, or headache-will be assessed weekly during the treatment phase (Weeks 4 to 7), also using 'yes' or 'no' responses.
Satisfaction with Treatment | Assessment timepoints: Week 8 (Visit 4/after completing the four-week treatment with active [a-tDCS], sham [s-tDCS], or duloxetine)
  Assessed using the Numeric Satisfaction with Treatment Scale (NSTS), ranging from 0 (not at all satisfied) to 10 (extremely satisfied).
Global Cognitive Function (MoCA) | Assessment timepoints: Baseline; Week 8 (Visit 4/after completing the four-week treatment with active [a-tDCS], sham [s-tDCS], or duloxetine)
  Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA), a screening tool for global cognition. Scores range from 0 to 30, with higher scores indicating better cognitive performance. A score below 26 is suggestive of cognitive impairment
Attention and Working Memory (Digit Span - WAIS-III) | Assessment timepoints: Baseline; Week 8 (Visit 4/after completing the four-week treatment with active [a-tDCS], sham [s-tDCS], or duloxetine)
  Attention and working memory will be assessed using the Digit Span subtest of the WAIS-III. The total score is based on correct forward and backward digit recall, with higher scores indicating better performance.
Processing Speed (Symbol Search - WAIS-III) | Assessment timepoints: Baseline; Week 8 (Visit 4/after completing the four-week treatment with active [a-tDCS], sham [s-tDCS], or duloxetine)
  Processing speed will be assessed using the Symbol Search subtest of the WAIS-III. The outcome is a scaled score ranging from 1 to 19, with higher scores indicating faster processing.
Inhibitory Control (Stop Signal Task) | Assessment timepoints: Baseline; Week 8 (Visit 4/after completing the four-week treatment with active [a-tDCS], sham [s-tDCS], or duloxetine)
  Inhibitory control will be assessed using the Stop Signal Task. The primary outcome is Stop Signal Reaction Time (SSRT), measured in milliseconds. Lower reaction times indicate better inhibitory control.
Cognitive Flexibility (Trail Making Test A and B) | Assessment timepoints: Baseline; Week 8 (Visit 4/after completing the four-week treatment with active [a-tDCS], sham [s-tDCS], or duloxetine)
  Executive function and cognitive flexibility will be assessed using the Trail Making Test Parts A and B. The outcome is total time to completion in seconds. Longer completion times indicate worse performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon request at wcaumo@hcpa.edu.br after 6 months of publication Data available: Yes. When available: With publication. Data types: Deidentified participant data, Data dictionary. Additional Information Who can access the data: Anyone requesting the data. Types of analyses: For any purpose. Mechanisms of data availability: Without investigator support.
Supporting Information: Study Protocol, SAP
Time Frame: When available: With publication of primary outcomes
Access Criteria: Data will be available upon request at wcaumo@hcpa.edu.br after 6 months of publication

REFERENCES:
- [Result] Yousefi Soorani L, Shafiei Bafti B, Homam SM, Abbasloo Z, Taghizadeh Zanooghi H. Hypogene enrichment in Miduk porphyry copper ore deposit, Iran. Sci Rep. 2022 Nov 9;12(1):19133. doi: 10.1038/s41598-022-23501-5. PMID 36352022
- [Result] Jornada MND, Antunes LC, Alves C, Torres ILS, Fregni F, S Sanches PR, P Silva D Jr, Caumo W. Impact of multiple-session home-based transcranial direct current stimulation (M-HB-tDCS) on eating behavior in fibromyalgia: A factorial randomized clinical trial. Brain Stimul. 2024 Mar-Apr;17(2):152-162. doi: 10.1016/j.brs.2024.02.001. Epub 2024 Feb 8. PMID 38336340
- [Result] Fregni F, El-Hagrassy MM, Pacheco-Barrios K, Carvalho S, Leite J, Simis M, Brunelin J, Nakamura-Palacios EM, Marangolo P, Venkatasubramanian G, San-Juan D, Caumo W, Bikson M, Brunoni AR; Neuromodulation Center Working Group. Evidence-Based Guidelines and Secondary Meta-Analysis for the Use of Transcranial Direct Current Stimulation in Neurological and Psychiatric Disorders. Int J Neuropsychopharmacol. 2021 Apr 21;24(4):256-313. doi: 10.1093/ijnp/pyaa051. PMID 32710772
- [Result] Caumo W, Lopes Ramos R, Vicuna Serrano P, da Silveira Alves CF, Medeiros L, Ramalho L, Tomeddi R, Bruck S, Boher L, Sanches PRS, Silva DP Jr, Ls Torres I, Fregni F. Efficacy of Home-Based Transcranial Direct Current Stimulation Over the Primary Motor Cortex and Dorsolateral Prefrontal Cortex in the Disability Due to Pain in Fibromyalgia: A Factorial Sham-Randomized Clinical Study. J Pain. 2024 Feb;25(2):376-392. doi: 10.1016/j.jpain.2023.09.001. Epub 2023 Sep 7. PMID 37689323
- [Result] Caumo W, Deitos A, Carvalho S, Leite J, Carvalho F, Dussan-Sarria JA, Lopes Tarrago Mda G, Souza A, Torres IL, Fregni F. Motor Cortex Excitability and BDNF Levels in Chronic Musculoskeletal Pain According to Structural Pathology. Front Hum Neurosci. 2016 Jul 15;10:357. doi: 10.3389/fnhum.2016.00357. eCollection 2016. PMID 27471458
- [Result] Caumo W, Alves RL, Vicuna P, Alves CFDS, Ramalho L, Sanches PRS, Silva DP, da Silva Torres IL, Fregni F. Impact of Bifrontal Home-Based Transcranial Direct Current Stimulation in Pain Catastrophizing and Disability due to Pain in Fibromyalgia: A Randomized, Double-Blind Sham-Controlled Study. J Pain. 2022 Apr;23(4):641-656. doi: 10.1016/j.jpain.2021.11.002. Epub 2021 Nov 13. PMID 34785366
- [Result] Brietzke AP, Zortea M, Carvalho F, Sanches PRS, Silva DPJ, Torres ILDS, Fregni F, Caumo W. Large Treatment Effect With Extended Home-Based Transcranial Direct Current Stimulation Over Dorsolateral Prefrontal Cortex in Fibromyalgia: A Proof of Concept Sham-Randomized Clinical Study. J Pain. 2020 Jan-Feb;21(1-2):212-224. doi: 10.1016/j.jpain.2019.06.013. Epub 2019 Jul 26. PMID 31356985

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-03): https://cdn.clinicaltrials.gov/large-docs/39/NCT07203339/Prot_SAP_000.pdf